CLINICAL TRIAL: NCT00532701
Title: Peginterferon Alfa-2a Plus Ribavirin in Patients With Genotype 2 Chronic Hepatitis C: A Randomized Study of Treatment Duration and Ribavirin Dose Stratified by Rapid Virologic Response
Brief Title: Peginterferon Alfa-2a and Ribavirin for Genotype 2 Chronic Hepatitis C: Duration and Ribavirin Dose Stratified by RVR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200709014M
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Genotype; Interferon; Ribavirin; Genotype 2; Peginterferon
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Peg-IFN + WB RBV for 16 weeks (Active Comparator): Weight-based ribavirin (1000-1200 mg/day) from weeks 1-16 in patients with RVR
  Interventions: Drug: Peg-IFN + WB RBV for 16 weeks
- Peg-IFN + LD RBV for 16 weeks (Active Comparator): Weight-based ribavirin (1000-1200 mg/day) from weeks 1-6, and then low dose ribavirin (800 mg/day) from weeks 6-16 in patients with RVR
  Interventions: Drug: Peg-IFN + LD RBV for 16 weeks
- Peg-IFN + WB RBV for 24 weeks (Active Comparator): Weight-based ribavirin (1000-1200 mg/day) from weeks 1-24 in patients without RVR
  Interventions: Drug: Peg-IFN + WB RBV for 24 weeks
- Peg-IFN + WB RBV for 48 weeks (Active Comparator): Weight-based ribavirin (1000-1200 mg/day) from weeks 1-48 in patients without RVR
  Interventions: Drug: Peg-IFN + WB RBV for 48 weeks
- Peg-IFN + LD RBV for 24 weeks (Active Comparator): Low dose ribavirin (800 mg/day) from weeks 1-24 in patients with or without RVR
  Interventions: Drug: Peg-IFN + LD RBV for 24 weeks

INTERVENTIONS:
Drug: Peg-IFN + WB RBV for 16 weeks — 1. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day (< 75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) from weeks 1-4
  2. Rapid virologic response (RVR) at week 4 of therapy: achieved
  3. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day (< 75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) from weeks 5-16
  Other Names: Pegasys plus Copegus
  Arms: Peg-IFN + WB RBV for 16 weeks
Drug: Peg-IFN + LD RBV for 16 weeks — 1. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day (< 75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) from weeks 1-6
  2. Rapid virologic response (RVR) at week 4 of therapy: achieved
  3. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 800 mg/day from weeks 6-16
  Other Names: Pegasys plus Copegus
  Arms: Peg-IFN + LD RBV for 16 weeks
Drug: Peg-IFN + WB RBV for 24 weeks — 1. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day (< 75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) from weeks 1-4
  2. Rapid virologic response (RVR) at week 4 of therapy: not achieved
  3. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day from weeks 5-24
  Other Names: Pegasys plus Copegus
  Arms: Peg-IFN + WB RBV for 24 weeks
Drug: Peg-IFN + WB RBV for 48 weeks — 1. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day (< 75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) from weeks 1-4
  2. Rapid virologic response (RVR) at week 4 of therapy: not achieved
  3. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 1000-1200 mg/day from weeks 5-48
  Other Names: Pegasys plus Copegus
  Arms: Peg-IFN + WB RBV for 48 weeks
Drug: Peg-IFN + LD RBV for 24 weeks — 1. Peginterferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 180 ug/week plus ribavirin (Copegus, Hoffman-LaRoche) 800 mg/day from weeks 1-24
  2. Rapid virologic response (RVR) at week 4 of therapy: both achieved and not achieved
  Other Names: Pegasys plus Copegus
  Arms: Peg-IFN + LD RBV for 24 weeks

SUMMARY:
Treatment with peginterferon plus daily low dose (800 mg) or weight-based ribavirin (800-1400 mg) for 24 to 48 weeks has achieved 70-93% sustained virologic response (SVR) rates in patients with genotype 2 or 3 chronic hepatitis C (CHC). Recently, a large randomized study has shown that patients with genotype 2 or 3 CHC have comparable SVR rates for those who received peginterferon for 24 or 48 weeks, and who received daily low dose (800 mg) or standard dose (1000-1200 mg) ribavirin. Therefore, the currently recommended treatment for these patients is 24 weeks of peginterferon plus low dose ribavirin. Because of the high response rates, several studies have shown that when these patients had rapid virologic response (RVR), defined as undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) levels, at week 4 of peginterferon plus weight-based ribavirin, 12-16 weeks of treatment could have 82-94% SVR rates. However, treatment with peginterferon plus low dose ribavirin for 24 weeks showed significantly higher SVR rates than that for 16 weeks (85% versus 79%) in these patients who achieved RVR. While studies showed concordant results in SVR rates for patients with genotype 3 CHC who received peginterferon plus low dose or weight-based ribavirin for 16 or 24 weeks, the SVR rates stratified by RVR showed great differences in patients with genotype 2 CHC who received such treatment. Currently, there are no studies on the direct comparison of low dose versus weight-based ribavirin, and of 16 to 24 weeks of treatment stratified by RVR for patients with genotype 2 CHC. The investigators aimed to conduct a randomized trial to determine the optimal ribavirin dose and treatment duration of peginterferon plus ribavirin for patients with genotype 2 CHC based on RVR studies.

DETAILED DESCRIPTION:
Treatment with peginterferon plus daily low dose (800 mg) or weight-based ribavirin (800-1400 mg) for 24 to 48 weeks has achieved 70-93% sustained virologic response (SVR) rates in patients with genotype 2 or 3 chronic hepatitis C (CHC). Recently, a large randomized study has shown that patients with genotype 2 or 3 CHC have comparable SVR rates for those who received peginterferon for 24 or 48 weeks, and who received daily low dose (800 mg) or standard dose (1000-1200 mg) ribavirin. Therefore, the currently recommended treatment for these patients is 24 weeks of peginterferon plus low dose ribavirin. Because of the high response rates, several studies have shown that when these patients had rapid virologic response (RVR), defined as undetectable hepatitis C virus (HCV) RNA levels, at week 4 of peginterferon plus weight-based ribavirin, 12-16 weeks of treatment could have 82-94% SVR rates. However, treatment with peginterferon plus low dose ribavirin for 24 weeks showed significantly higher SVR rates than that for 16 weeks (85% vs. 79%) in these patients who achieved RVR. While studies showed concordant results in SVR rates for patients with genotype 3 CHC who received peginterferon plus low dose or weight-based ribavirin for 16 or 24 weeks, the SVR rates stratified by RVR showed great differences in patients with genotype 2 CHC who received such treatment. Currently, there are no studies on the direct comparison of low dose versus weight-based ribavirin, and of 16 to 24 weeks of treatment stratified by RVR for patients with genotype 2 CHC. We aimed to conduct a randomized trial to determine the optimal ribavirin dose and treatment duration of peginterferon plus ribavirin for patients with genotype 2 CHC based on RVR studies.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Age older than 18 years old
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Taqman HCV Monitor v2.0, Roche Diagnostics) with dynamic range 25 ~ 391000000 IU/ml
* HCV genotype 2 (Inno-LiPA HCV II, Innogenetics, Ghent, Belgium)
* Serum alanine aminotransferase levels above the upper limit of normal with 6 months of enrollment
* A liver biopsy consistent with the diagnosis of chronic hepatitis C

Exclusion Criteria:

* Anemia (hemoglobin < 13 grams per deciliter for men and < 12 grams per deciliter for women)
* Neutropenia (neutrophil count < 1,500 per cubic milliliter)
* Thrombocytopenia (platelets < 90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic alcohol abuse (daily consumption > 20 grams per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to use contraception
* Unwilling to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2007-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 1.5 year

SECONDARY OUTCOMES:
Histologic response (HR) | 1.5 year
Biochemical response (BR) | 1.5

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, MD, PhD, Principal Investigator — National Taiwan University Hospital; Ding-Shinn Chen, MD, Principal Investigator — National Taiwan University Hospital; Ming-Yang Lai, MD, PhD, Principal Investigator — National Taiwan University Hospital; Pei-Jer Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital; Chun-Jen Liu, MD, PhD, Principal Investigator — National Taiwan University Hospital; Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Chih-Lin Lin, MD, Principal Investigator — Taipei City Hospital, Ren-Ai Branch; Cheng-Chao Liang, MD, Principal Investigator — Far Eastern Memorial Hospital; Ching-Sheng Hsu, MD, Principal Investigator — Buddhist Xindian Tzu Chi General Hospital; Sheng-Shun Yang, MD, Principal Investigator — Taichung Veterans General Hospital; Chia-Chi Wang, MD, Principal Investigator — Buddhist Xindian Tzu Chi General Hospital; Tai-Chung Tseng, MD, Principal Investigator — Buddhist Xindian Tzu Chi General Hospital; Ming-Lung Yu, MD, PhD, Principal Investigator — Kaohsiung Medical University; Wan-Long Chuang, MD, PhD, Principal Investigator — Kaohsiung Medical University; Chia-Yen Dai, MD, Ms, Principal Investigator — Kaohsiung Municipal Hsiao-Kang Hospital; Jee-Fu Huang, MD, Principal Investigator — Kaohsiung Municipal Hsiao-Kang Hospital; Chang-Fu Chiu, MD, Principal Investigator — Paochien Hospital
Locations (9):
- Taiwan (9):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Kaohsiung Medical University, Kaohsiung City
  - Kaohsiung Municipal Hsiao-Kang Hospital, Kaohsiung City
  - Paochien Hospital, Pingtung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Buddhist Xindian Tzu Chi General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Ren-Ai Branch, Taipei Municipal Hospital, Taipei

REFERENCES:
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] Zeuzem S, Hultcrantz R, Bourliere M, Goeser T, Marcellin P, Sanchez-Tapias J, Sarrazin C, Harvey J, Brass C, Albrecht J. Peginterferon alfa-2b plus ribavirin for treatment of chronic hepatitis C in previously untreated patients infected with HCV genotypes 2 or 3. J Hepatol. 2004 Jun;40(6):993-9. doi: 10.1016/j.jhep.2004.02.007. PMID 15158341
- [Background] Shiffman ML, Suter F, Bacon BR, Nelson D, Harley H, Sola R, Shafran SD, Barange K, Lin A, Soman A, Zeuzem S; ACCELERATE Investigators. Peginterferon alfa-2a and ribavirin for 16 or 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2007 Jul 12;357(2):124-34. doi: 10.1056/NEJMoa066403. PMID 17625124
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920
- [Background] Dalgard O, Bjoro K, Hellum KB, Myrvang B, Ritland S, Skaug K, Raknerud N, Bell H. Treatment with pegylated interferon and ribavarin in HCV infection with genotype 2 or 3 for 14 weeks: a pilot study. Hepatology. 2004 Dec;40(6):1260-5. doi: 10.1002/hep.20467. PMID 15558712
- [Background] von Wagner M, Huber M, Berg T, Hinrichsen H, Rasenack J, Heintges T, Bergk A, Bernsmeier C, Haussinger D, Herrmann E, Zeuzem S. Peginterferon-alpha-2a (40KD) and ribavirin for 16 or 24 weeks in patients with genotype 2 or 3 chronic hepatitis C. Gastroenterology. 2005 Aug;129(2):522-7. doi: 10.1016/j.gastro.2005.05.008. PMID 16083709
- [Background] Mangia A, Santoro R, Minerva N, Ricci GL, Carretta V, Persico M, Vinelli F, Scotto G, Bacca D, Annese M, Romano M, Zechini F, Sogari F, Spirito F, Andriulli A. Peginterferon alfa-2b and ribavirin for 12 vs. 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2005 Jun 23;352(25):2609-17. doi: 10.1056/NEJMoa042608. PMID 15972867
- [Background] Yu ML, Dai CY, Huang JF, Hou NJ, Lee LP, Hsieh MY, Chiu CF, Lin ZY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL. A randomised study of peginterferon and ribavirin for 16 versus 24 weeks in patients with genotype 2 chronic hepatitis C. Gut. 2007 Apr;56(4):553-9. doi: 10.1136/gut.2006.102558. Epub 2006 Sep 6. PMID 16956917
- [Derived] Liu CH, Huang CF, Liu CJ, Dai CY, Huang JF, Lin JW, Liang CC, Yang SS, Lin CL, Su TH, Yang HC, Chen PJ, Chen DS, Chuang WL, Kao JH, Yu ML. Peginterferon plus weight-based ribavirin for treatment-naive hepatitis C virus genotype 2 patients not achieving rapid virologic response: a randomized trial. Sci Rep. 2015 Jul 1;5:11710. doi: 10.1038/srep11710. PMID 26130141